CLINICAL TRIAL: NCT01520246
Title: Signaling in Tumorigenesis and Immunity
Brief Title: Gene Expression in Samples From Patients With T-Cell Acute Lymphoblastic Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AALL12B2; COG-AALL12B2 (Other: Children's Oncology Group); CDR0000723902 (Other: clinicaltrials.gov); AALL12B2 (Other: COG); NCI-2012-00241 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-01-26; First posted 2012-01-27 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Leukemia; Lymphoma
Keywords: adult acute lymphoblastic leukemia; childhood acute lymphoblastic leukemia; adult T-cell leukemia/lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — Gene Expression Profiling

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — tissue, blood, and bodily fluids
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: gene expression analysis
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood and tissue from patients with cancer in the laboratory may help doctors identify and learn more about biomarkers related to cancer. It may also help doctors find better ways to treat cancer.

PURPOSE: This research trial studies gene expression in samples from patients with T-cell acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* To test whether the tumor suppressor candidate gene PDLIM2 is downregulated in human cancers such as T-cell acute lymphoblastic leukemia (T-ALL) and to use the human T-lymphotropic virus 1 (HTLV-1)-mediated in vitro transformation of human T cells as control.

OUTLINE: Previously collected cancer and control tissues are analyzed for the expression patterns of PDLIM2 and other control genes. Human T-cells isolated from human blood are also co-cultured with HTLV-1-transformed T-cell lines.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Specimens (e.g., tissue, blood, and bodily fluids) of various cancer cells and or tissues from de-identified patients such as T-cell acute lymphoblastic leukemia (T-ALL)
* Normal control tissue

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients With T-Cell Acute Lymphoblastic Leukemia
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2012-01; Primary Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
PDLIM2 expression patterns in cancer and control tissues
8-week survival of human T-cell co-cultured with HTLV-1-transformed T-cell lines

CONTACTS AND LOCATIONS:
Overall Officials: Gutian Xiao, MD, Principal Investigator — University of Pittsburgh